CLINICAL TRIAL: NCT07398430
Title: Metabolic Characteristics Analysis and Precise Prognostic Model Establishment for Patients With Acute Coronary Syndrome Complicated With Obstructive Sleep Apnea
Brief Title: Metabolic Characteristics and Prognostic Model of Acute Coronary Syndrome Complicated With Obstructive Sleep Apnea
Acronym: OSA-ACS-Met
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, WeiGong, Deputy Director, Beijing Hospital
Other Study IDs: 2025BJYYEC-KY309-02
Record Dates: First submitted 2026-02-04; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disordered Breathing (SDB)
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biological Sample Collection — Collection of blood, urine, and stool samples for metabolomics analysis.

SUMMARY:
Obstructive sleep apnea (OSA) significantly increases the risk of cardiovascular events in patients with acute coronary syndrome (ACS), yet the underlying metabolic mechanisms remain unclear. This study aims to analyze the metabolic characteristics of ACS patients with OSA using metabolomics based on a prospective cohort. The study intends to construct an artificial intelligence-based risk stratification model to improve prognosis prediction and facilitate precision medicine for this population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years.
* Diagnosed with ACS, including ST-segment elevation myocardial infarction, non-ST-segment elevation myocardial infarction, and unstable angina.
* Willing to participate and sign the informed consent form.

Exclusion Criteria:

* Cardiogenic shock or cardiac arrest.
* Central sleep apnea or other types of sleep disordered breathing.
* Previous or current treatment with continuous positive airway pressure.
* Inability to complete polysomnography or invalid data.
* Malignancy or life expectancy < 1 year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients diagnosed with ACS at Beijing Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 12 Months

IPD SHARING:
Plan to Share IPD: No